CLINICAL TRIAL: NCT02321241
Title: A retrospecTive and Prospective Non-Interventional Study to Assess the Clinical pracTice in Real Life for Patients With Wet AMD Refractory to raNibizumab and Switching to Aflibercept
Brief Title: Real Life of Aflibercept in France in Patients Refractory to Ranibizumab: Observational Study in Wet AMD
Acronym: TITAN
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 17405; EY1413FR (Other: company internal)
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Wet Macular Degeneration
Keywords: Wet-AMD; Refractory patients to ranibizumab; Real life; Switch; Aflibercept
MeSH Terms: conditions — Wet Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: According to the recommendations of the Summary of Products Characteristics (SmPC) Administration by intravitreal injection
  Interventions: Drug: Aflibercept (EYLEA, BAY-86-5321)

INTERVENTIONS:
Drug: Aflibercept (EYLEA, BAY-86-5321) — 1. st year: 3 monthly injections followed by 1 injection every two months
  2. nd year and following: injection according the visual and anatomical results observed the 1st year

SUMMARY:
The aim of the TITAN study is to describe the clinical practices of a cohort of patients with wAMD refractory to ranibizumab (persistence of intra-retinal and/or subretinal fluid) who switch to aflibercept after less than 12 months of ranibizumab treatment.

The study will be conducted in real-life conditions and will allow describing conditions of use of aflibercept in patients refractory to ranibizumab

DETAILED DESCRIPTION:
The study is both retrsopective and prospective to collect local real life data on patients under routine treatment.

The observation periods starts on January 2014. Patients who initiated a treatment by Aflibercept between the 1st of january 2014 and the 31 December 2015 will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman > 18 years old
* Patient with wAMD previously treated with ranibizumab (for less than 12 months before initiation of Aflibercept)
* Refractory to ranibizumab (defined by persistent fluid despite a treatment conducted according to the HAS French recommendations with at least 3 loading doses injections)
* Patient who switched to aflibercept (Eylea) between 1st of January 2014 and 30th June 2015
* Written informed consent given

Exclusion Criteria:

* Patient who do not meet the local indication criteria for aflibercept treatment. Contraindications listed in the local SmPC (Summary of Product Characteristics) have to be considered
* Recurrent patients with wAMD previously treated with ranibizumab and switched to aflibercept because of a high recurrence rate (recurrent patients described by Yonegawa et al.in AJO (American Journal of Ophthalmology )2013= exudation suppressed but high rate of injections)
* Patient who have been previously treated by any macular laser Visudyne/PD (Photodynamic therapy)
* Patient with a Visual Acuity (VA) <1/10
* Patient with Fibrosis involving Macula
* Patient with atrophic AMD
* Patient with any other retinal disease as myopia, diabetic retinopathy, diabetic macular oedema,chorioretinal anastomosis (CRA),, angioid streaks
* Patients taking part in an interventional study at the time of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of wAMD refractory to ranibizumab (persistence of fluid) who started a treatment with Anti VEGF (Aflibercept) may be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-08-18 (Actual)

PRIMARY OUTCOMES:
Treatment success rate (defined as a gain of at least 1 letter in BCVA and/or a diminution of CRT (expressed in µm)) | Between initial visit and 12 month follow up visit
  The 12 month follow up visit is the visit 12 month after the first injection of aflibercept

SECONDARY OUTCOMES:
Proportion of patients whose BCVA increases by ≥ 0 letter, ≥ 5 letters, ≥ 10 letters, ≥15 letters | Between initial visit and up to 1 year maximum
  The end of study visit is the visit 12 month after the first injection of aflibercept or after last follow up visit when the patient drop out the study whichever apply..
Proportion of patients with less than 15 letters loss | Between initial visit and up to 1 year maximum
Proportion of patients with dry-OCT | Between initial visit and up to 1 year maximum
Mean duration of treatment with ranibizumab before initiation of aflibercept | Between initial visit and up to 1 year maximum
Mean change in Central retinal thickness in µm (OCT) | Between initial visit and up to 1 year maximum

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, France

REFERENCES:
- [Derived] Razavi S, Kodjikian L, Giocanti-Auregan A, Dufour I, Souied E. Efficacy and safety of intravitreal aflibercept in ranibizumab-refractory patients with neovascular age-related macular degeneration. BMC Ophthalmol. 2021 Feb 17;21(1):90. doi: 10.1186/s12886-021-01841-6. PMID 33596867